CLINICAL TRIAL: NCT04798989
Title: A Phase 2a Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CY6463 When Administered to Participants With Alzheimer's Disease and Vascular Pathology
Brief Title: A Study of the Effects of CY6463 in Participants With Alzheimer's Disease With Vascular Pathology
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C6463-202
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease With Vascular Pathology
Keywords: Alzheimer's disease; AD; ADv; CY6463; Subcortical small-vessel disease; Elderly; 60 and older; Probable AD dementia; Vascular dementia; Mixed dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CY6463 (Experimental): CY6463 once daily (QD) for approximately 87 sequential days.
  Interventions: Drug: CY6463
- Placebo (Placebo Comparator): Placebo QD for approximately 87 sequential days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CY6463 — CY6463 Oral Tablet
  Other Names: IW-6463; zagociguat
  Arms: CY6463
Drug: Placebo — Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
This study is being conducted to test the safety, tolerability, and pharmacokinetics of the investigational drug CY6463 compared with placebo in individuals who are aged 60 years or older and have Alzheimer's disease (AD) along with common cardiovascular risk factors.

DETAILED DESCRIPTION:
CY6463 is an investigational drug being developed as a symptomatic and potentially disease-modifying therapy for Alzheimer's disease (AD) and other serious central nervous system disorders. As a soluble guanylate cyclase (sGC) stimulator, CY6463 can cross the blood-brain barrier and boosts the activity of the nitric oxide-soluble guanylate cyclase-cyclic guanosine monophosphate (NO-sGC-cGMP) pathway. This signaling pathway is important in many aspects of brain health, including in the control of blood flow in the brain, how brain cells use energy, and how those cells communicate with one another. Impairment of this pathway is a critical part of the origin of many neurodegenerative diseases that can cause a loss of brain function including memory and decision-making abilities. There are clear links between disrupted NO signaling and impaired brain function in patients with AD and vascular pathology (ADv). ("Vascular pathology" refers to abnormalities of the blood vessels that are more likely to occur when a person has cardiovascular risk factors like high blood pressure, diabetes, and/or obesity.) It is hypothesized that CY6463 may help patients with ADv maintain or recover some of their original cognitive function.

In this study, participants will be randomized to receive approximately 87 sequential days (~3 months) of study drug (CY6463 or placebo) once daily (QD) and will complete 7 scheduled site visits over the course of the study, from Screening through Follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to the performance of any protocol-specified procedure or, if unable to provide informed consent due to cognitive status, provides assent to participate, with a legally authorized representative (LAR) providing written informed consent on behalf of the participant.
2. 60 years of age or older
3. Meets core clinical criteria for probable AD dementia according to the 2011 National Institute on Aging-Alzheimer's Associated guidelines. Can be based on medical history.
4. Mini-Mental State Examination (MMSE) score of 20 to 26 (inclusive)
5. Confirmation of AD pathophysiology
6. At least 2 cardiovascular risk factors per protocol criteria
7. Magnetic resonance imaging (MRI) scan (existing MRI obtained ≤6 months before Screening is acceptable) findings of mild-to-moderate subcortical small-vessel disease
8. If receiving concomitant or chronic medication(s), has had no change for ≥4 weeks before study drug initiation and has no plans to alter the regimen(s) during the study
9. If male, agrees to refrain from donating sperm from the Screening visit through 90 days after taking the final study drug dose
10. If male, agrees to use protocol-specified, effective contraception methods from the signing of the informed consent form (ICF) until ≥90 days after taking the final study drug dose.
11. If female, is postmenopausal/not of reproductive potential defined per protocol
12. Agrees to the study procedures, including undergoing lumbar puncture for cerebrospinal fluid (CSF) samples

Exclusion Criteria:

1. Severe visual, auditory, social, or cognitive impairment
2. Dementia-related disorder other than AD or vascular dementia (eg, Parkinson's disease, Huntington's disease, frontotemporal dementia, schizophrenia, Lewy body dementia)
3. Symptomatic large-vessel disease, symptomatic carotid artery disease, large vessel infarcts, or strategic lacunar infarcts or infarcts>15 mm
4. History of significant central nervous system (CNS) trauma that has affected brain function
5. Low blood pressure (BP), defined as systolic BP ≤90 mmHg or diastolic BP ≤60 mmHg.
6. Orthostatic hypotension.
7. Unable to undergo MRI
8. Unable to undergo lumbar puncture procedure
9. Unable to participate in electroencephalography (EEG) protocol due to hearing impairment or inability to tolerate EEG cap or headphones
10. Uncontrolled or unstable chronic disease
11. Kidney impairment requiring dialysis; history of renal transplant
12. Needs continuous direct medical care and nursing supervision.
13. Family history of short QT syndrome or long QT syndrome
14. Clinically significant cardiac involvement
15. History of cancer. Exceptions: localized cutaneous basal or squamous cell carcinoma in the last 5 years, low-grade localized prostate/cervical cancers, or previous localized prostate/cervical cancers that have a low likelihood of recurrence
16. Is not suited for study participation in the clinical judgment of the investigator

Additional inclusion and exclusion criteria apply, per protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Tisento Therapeutics
Locations (5):
- United States (5):
  - Clinical Endpoints, Scottsdale, Arizona
  - Optimus U Corp, Miami, Florida
  - Hawaii Pacific Neurosciences, LLC, Honolulu, Hawaii
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either CY6463 or placebo.
Groups:
- Placebo: Placebo once daily (QD) for approximately 87 sequential days.
- CY6463: CY6463 QD for approximately 87 sequential days.
Period: Overall Study
Arm/Group | Placebo | CY6463
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CY6463 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  White | 3 | 4 | 7
  Black or African American | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs) From Study Drug Initiation Through Follow-up
Description: TEAE is defined as an adverse event with an onset that occurs after receiving the study drug, until the end of the Follow-up period
Time Frame: From first dose of study treatment through ~14 (±4) days after the final dose
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CY6463
Number analyzed (Participants) | 6 | 6
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: From informed consent through ~14 (±4) days after the final dose. (Dosing ranged from 84 to 90 days for placebo and 85 to 91 days for CY6463).
Arm/Group | Placebo | CY6463
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | CY6463 (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04798989/Prot_SAP_000.pdf